CLINICAL TRIAL: NCT07339423
Title: Efficacy and Safety of NNC0487-0111 s.c. Once-weekly in Participants With Obesity (AMAZE 1)
Brief Title: AMAZE 1: A Research Study Investigating How Well the Medicine NNC0487-0111 Helps People With Excess Body Weight Lose Weight
Acronym: AMAZE 1
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9490-8021; U1111-1313-6262 (Other: World Health Organization (WHO)); 2024-520440-42 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2026-01-13; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC0487-0111 (Experimental): Participants will be randomized to receive 1 out of 4 different dose levels subcutaneously once weekly as an adjunct to a reduced-calorie diet and increased physical activity.
  Interventions: Drug: NNC0487-0111
- Placebo (Placebo Comparator): Participants will receive placebo matched to NNC0487-0111 subcutaneously once weekly as an adjunct to a reduced-calorie diet and increased physical activity.
  Interventions: Drug: Placebo (matched to NNC0487-0111)

INTERVENTIONS:
Drug: NNC0487-0111 — NNC0487-0111 will be administered subcutaneously using PDS290 pre-filled pen-injectors to one of the body parts: thigh, abdomen or upper arm.
  Arms: NNC0487-0111
Drug: Placebo (matched to NNC0487-0111) — Placebo matched to NNC0487-0111 will be administered subcutaneously using PDS290 pre-filled pen-injectors to one of the body parts: thigh, abdomen or upper arm.
  Arms: Placebo

SUMMARY:
The purpose of this clinical study is to find out if NNC0487-0111 is safe and effective for treating people who have excess body weight. There are 2 study treatments in this study taken as injections under the skin once a week. Participants will either get NNC0487-0111 (the treatment being tested) or Placebo (a treatment that has no active medicine in it). Which treatment participants get is decided by chance.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female (sex at birth).
* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* History of at least one self-reported unsuccessful dietary effort to lose body weight.

Key Exclusion Criteria:

* HbA1c ≥ 6.5% (48 millimole per mole [mmol/mol]) as measured by the central laboratory at screening.
* History of type 1 or type 2 diabetes mellitus as declared by the participant or reported in the medical records.
* Treatment with glucagon-like-peptide-1 (GLP-1) receptor agonists (RA), dual GLP-1/gastric inhibitory peptide (GIP) RAs (or any other GLP-1 based treatment) or amylin analogues before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2029-06-26 (Estimated); Study Completion 2029-08-21 (Estimated)

PRIMARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to week 84
  Measured as percentage of body weight.

SECONDARY OUTCOMES:
Change in waist circumference | From baseline (week 0) to week 84 and week 136
  Measured as centimetre (cm).
Change in systolic blood pressure (SBP) | From baseline (week 0) to week 84 and week 136
  Measured as millimetre of mercury (mmHg).
Change in Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite-CT) physical function score | From baseline (week 0) to week 84 and week 136
  Measured as score on a scale. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. The physical function score ranges from 0-100.
Change in SF-36v2® Health Survey Acute (SF-36v2 Acute) physical functioning score | From baseline (week 0) to week 84 and week 136
  Measured as score on a scale. SF-36v2 Acute measures Health-Related Quality of Life (HRQOL). The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 Acute scores are norm-based scores, i.e. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation (SD) of 10. Higher scores indicate better functional health and well-being. The physical functioning ranges from 19.0 to 57.6.
Change in body weight | From baseline (week 0) to week 84 and week 136
  Measured as kilogram (kg).
Change in body mass index (BMI) | From baseline (week 0) to week 84 and week 136
  Measured as kilograms per meter squared (kg/m^2).
Change in IWQOL-Lite-CT physical composite score | From baseline (week 0) to week 84 and week 136
  Measured as score on a scale. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. The physical composite score ranges from 0-100.
Change in IWQOL-Lite-CT psychosocial composite score | From baseline (week 0) to week 84 and week 136
  Measured as score on a scale. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. The psychosocial composite score ranges from 0-100.
Change in IWQOL-Lite-CT total score | From baseline (week 0) to week 84 and week 136
  Measured as score on a scale. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. The total score ranges from 0-100.
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to week 84 and week 136
  Measured as percentage of HbA1c.
Change in fasting plasma glucose (FPG) | From baseline (week 0) to week 84 and week 136
  Measured as millimole per liter (mmol/L).
Ratio to baseline: change in fasting insulin | From baseline (week 0) to week 84 and week 136
  Measured as ratio.
Change in diastolic blood pressure (DBP) | From baseline (week 0) to week 84
  Measured as mmHg.
Ratio to baseline: change in total cholesterol | From baseline (week 0) to week 84 and week 136
  Measured as ratio.
Ratio to baseline: change in high-density lipoprotein (HDL) cholesterol | From baseline (week 0) to week 84 and week 136
  Measured as ratio.
Ratio to baseline: change in low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to week 84 and week 136
  Measured as ratio.
Ratio to baseline: change in very low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to week 84 and week 136
  Measured as ratio.
Ratio to baseline: change in non-HDL cholesterol | From baseline (week 0) to week 84 and week 136
  Measured as ratio.
Ratio to baseline: change in triglycerides | From baseline (week 0) to week 84 and week 136
  Measured as ratio.
Ratio to baseline: change in high-sensitivity C-reactive protein (hsCRP) | From baseline (week 0) to week 84 and week 136
  Measured as ratio.
Number of treatment emergent adverse events (TEAEs) | From baseline (week 0) to week 84 and week 140
  Measured as events.
Number of treatment emergent serious adverse events (TESAEs) | From baseline (week 0) to week 84 and week 140
  Measured as events.
Number of TEAEs leading to permanent treatment discontinuation | From baseline (week 0) to week 84 and week 140
  Measured as events.
Relative change in body weight | From baseline (week 0) to week 136
  Measured as % of body weight.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (72):
- United States (22):
  - South Broward Research LLC, Miramar, Florida
  - Clinical Neuroscience Solution, Orlando, Florida
  - Hope Clin Res & Wellness, Conyers, Georgia
  - Endeavor Health, Skokie, Illinois
  - Midwest Inst For Clin Res, Indianapolis, Indiana
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - New York Gastroenterology Associates, New York, New York
  - UNC Eastowne Medical Office, Chapel Hill, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Accellacare, Wilmington, North Carolina
  - UPA Ctr Weight and Eating Dis, Philadelphia, Pennsylvania
  - Clinical Res Collaborative, Cumberland, Rhode Island
  - Medical Uni of SC Charleston, Charleston, South Carolina
  - Coastal Carolina Research Ctr, North Charleston, South Carolina
  - Hillcrest Clinical Research, Simpsonville, South Carolina
  - Amarillo Medical Specialists, Amarillo, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - Care United Research, LLC, Forney, Texas
  - Washington Cntr Weight Mgmt, Arlington, Virginia
  - Health Res of Hampton Roads, Newport News, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Rainier Clin Res Ctr Inc, Renton, Washington
- Argentina (6):
  - Fundación CESIM, Santa Rosa, La Pampa Province
  - Centro Medico Dra. Laura Maffei e Investigacion Clínica Apli, Buenos Aires
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - Sanatorio Esperanza, Esperanza, Santa Fe
  - CIPADI, Godoy Cruz
  - Instituto de Investigaciones Clinicas San Nicolás, San Nicolás
- Australia (4):
  - Sydney Clinical Trials, Campbelltown, New South Wales
  - Sydney Cardiometabolic Centre, Liverpool, New South Wales
  - Hunter Diabetes Centre, Merewether, New South Wales
  - Heart of Australia, Chelmer, Queensland
- Belgium (6):
  - HUB - Hôpital Erasme, Brussels
  - UZA - UZ Antwerpen - Department of Endocrinology, Edegem
  - UZ Gent - Endocrinologie - Diabetologie, Ghent
  - UZ Leuven - Endocrinology, Leuven
  - MECLINAS, Mechelen
  - AZ Delta - Roeselare, Roeselare
- Canada (5):
  - C-endo Diab Endo Clin Calgery, Calgary, Alberta
  - Ocean West Research Clinic, Surrey, British Columbia
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Nova Scotia Hlth Halifax, Halifax, Nova Scotia
  - Milestone Research, London, Ontario
- Denmark (6):
  - Sanos Clinic - Gandrup, Gandrup
  - Steno Diabetes Center Nordjylland, Gistrup
  - Gentofte Hospital - Center for Klinisk Metabolisk Forskning, Hellerup
  - Hillerød Endokrinologisk amb. H0652, Hillerød
  - Hvidovre Hospital Endokrinologisk forsknings afsnit 159, Hvidovre
  - Sanos Clinic - Vejle, Vejle
- France (5):
  - HOPITAL EUROPEEN GEORGES POMPIDOU_Service de nutrition et diabétologie, Paris
  - HCL-HOPITAL LYON SUD_Service d'Endocrinologie-Diabète-Nutrition, Pierre-Bénite
  - CHU NANTES - HOPITAL NORD LAENNEC_Service d'Endocrinologie-Diabétologie-Nutrition, Saint-Herblain
  - CENTRE HOSPITALIER UNIVERSITAIRE DE TOULOUSE-HOPITAL RANGUEIL-Service de diabétologie et nutrition, Toulouse
  - Centre de Recherche Clinique Portes Du Sud, Vénissieux
- Germany (6):
  - Herz- und Diabeteszentrum NRW - Bad Oeynhausen, Bad Oeynhausen
  - Zentrum fuer klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - MVZ im Altstadt-Carree Fulda GmbH - Zentrum für klinische Studien, Fulda
  - SMO.MD GmbH - Zentrum für klinische Studien, Magdeburg
  - Institut für Diabetesforschung Osnabrück, Osnabrück
  - Forschungszentrum Ruhr KliFoCenter GmbH, Kahrmann, Witten
- United Kingdom (12):
  - Fowey River Practice, Fowey, Cornwall
  - The Adam Practice, Poole, Dorset
  - Pickering Medical Practice, Pickering, North Yorkshire
  - Crouch Oak Family Practice, Addlestone, Surrey
  - The Health Centre, Bradford-on-Avon
  - EMS Healthcare, Cheshire
  - HMC Health - Hounslow, Hounslow
  - Kiltearn Medical Centre, Nantwich
  - Knowle House Surgery, Plymouth
  - Clifton Medical Centre, Rotherham
  - Staploe Medical Centre, Soham
  - Albany House Medical Centre, Wellingborough

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com